CLINICAL TRIAL: NCT03801707
Title: An Open Label, Proof of Concept Study to Evaluate the Feasibility and Safety of Kidney Transplant From HCV Positive Donors Into HCV Negative Recipient
Brief Title: Utilization of Hepatitis C Positive Kidneys in Negative Recipients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Reem Daloul, Assistant Professor of Clinical Medicine, Transplant Nephrology, Ohio State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018H0499
Record Dates: First submitted 2019-01-09; First posted 2019-01-11 (Actual); Results first posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-08

CONDITIONS: Kidney Transplant; Hepatitis C; HCV
MeSH Terms: conditions — Hepatitis C | interventions — Sofosbuvir; velpatasvir; sofosbuvir-velpatasvir drug combination; glecaprevir; pibrentasvir; glecaprevir and pibrentasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention group (Experimental): kidney transplant recipients who receive kidney allograft from hepatitis C viremic donors followed by treatment with direct acting antiviral therapies.
  Interventions: Drug: Sofosbuvir / Velpatasvir Oral Tablet [Epclusa]; Drug: Glecaprevir/Pibrentasvir 100 MG-40 MG Oral Tablet [MAVYRET]

INTERVENTIONS:
Drug: Sofosbuvir / Velpatasvir Oral Tablet [Epclusa] — fixed dose combination medication once a day for 12 weeks for the treatment of hepatitis C
  Other Names: Epclusa
Drug: Glecaprevir/Pibrentasvir 100 MG-40 MG Oral Tablet [MAVYRET] — Three tablets once a day for 12 weeks for treatment of hepatitis C
  Other Names: Mavyret

SUMMARY:
To evaluate the safety and feasibility of transplanting kidneys from Hepatitis C virus (HCV) infected donors into recipients without HCV infection

DETAILED DESCRIPTION:
This will be an open label, prospective, interventional, proof of concept study to evaluate the feasibility and safety of kidney transplant from HCV positive donors into HCV negative recipients using treatment with pan-genotypic direct acting antiviral therapies (DAAS) for treatment of post-transplant HCV transmission

ELIGIBILITY:
Recipient Inclusion/Exclusion Criteria:

Inclusion Criteria:

* Adult age >18 years able to provide consent
* Lack of available living donor
* Calculated pre-transplant reactive panel (cPRA) of <80%
* Estimated post-transplant survival (EPTS) index >20% and <80%
* Negative pre-transplant human immunodeficiency virus (HIV), hepatitis C virus (HCV), and hepatitis B virus (HBV) serology and blood HCV polymerase chain reaction (PCR)
* No clinically significant pre-transplant liver disease

Exclusion Criteria:

* Living donor available
* Dialysis time >5 years
* Listing for multi-organ transplantation
* Active or recent history (<6 months) of alcohol abuse or substance abuse
* Clinically significant liver disease as determined by principal investigator
* History of hepatocarcinoma
* Pregnancy or lactation
* Refusal to accept blood transfusion
* HIV infection
* HCV pcr or antibody positive
* HBV infection

Donor Inclusion Criteria:

* Positive HCV PCR at time of donation
* Kidney donor profile index (KDPI)<85%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2019-03-22 (Actual); Primary Completion 2021-04-28 (Actual); Study Completion 2021-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Reem Daloul, MD, Principal Investigator — Ohio State University School of Biomedical Science: The Ohio State University College of Medicine
Locations (1):
- Brenda Cuson, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hart A, Smith JM, Skeans MA, Gustafson SK, Wilk AR, Robinson A, Wainright JL, Haynes CR, Snyder JJ, Kasiske BL, Israni AK. OPTN/SRTR 2016 Annual Data Report: Kidney. Am J Transplant. 2018 Jan;18 Suppl 1(Suppl 1):18-113. doi: 10.1111/ajt.14557. PMID 29292608
- [Background] Curry MP, O'Leary JG, Bzowej N, Muir AJ, Korenblat KM, Fenkel JM, Reddy KR, Lawitz E, Flamm SL, Schiano T, Teperman L, Fontana R, Schiff E, Fried M, Doehle B, An D, McNally J, Osinusi A, Brainard DM, McHutchison JG, Brown RS Jr, Charlton M; ASTRAL-4 Investigators. Sofosbuvir and Velpatasvir for HCV in Patients with Decompensated Cirrhosis. N Engl J Med. 2015 Dec 31;373(27):2618-28. doi: 10.1056/NEJMoa1512614. Epub 2015 Nov 16. PMID 26569658
- [Background] Feld JJ, Jacobson IM, Hezode C, Asselah T, Ruane PJ, Gruener N, Abergel A, Mangia A, Lai CL, Chan HL, Mazzotta F, Moreno C, Yoshida E, Shafran SD, Towner WJ, Tran TT, McNally J, Osinusi A, Svarovskaia E, Zhu Y, Brainard DM, McHutchison JG, Agarwal K, Zeuzem S; ASTRAL-1 Investigators. Sofosbuvir and Velpatasvir for HCV Genotype 1, 2, 4, 5, and 6 Infection. N Engl J Med. 2015 Dec 31;373(27):2599-607. doi: 10.1056/NEJMoa1512610. Epub 2015 Nov 16. PMID 26571066
- [Background] Feld JJ, Moreno C, Trinh R, Tam E, Bourgeois S, Horsmans Y, Elkhashab M, Bernstein DE, Younes Z, Reindollar RW, Larsen L, Fu B, Howieson K, Polepally AR, Pangerl A, Shulman NS, Poordad F. Sustained virologic response of 100% in HCV genotype 1b patients with cirrhosis receiving ombitasvir/paritaprevir/r and dasabuvir for 12weeks. J Hepatol. 2016 Feb;64(2):301-307. doi: 10.1016/j.jhep.2015.10.005. Epub 2015 Oct 22. PMID 26476290
- [Background] Foster GR, Afdhal N, Roberts SK, Brau N, Gane EJ, Pianko S, Lawitz E, Thompson A, Shiffman ML, Cooper C, Towner WJ, Conway B, Ruane P, Bourliere M, Asselah T, Berg T, Zeuzem S, Rosenberg W, Agarwal K, Stedman CA, Mo H, Dvory-Sobol H, Han L, Wang J, McNally J, Osinusi A, Brainard DM, McHutchison JG, Mazzotta F, Tran TT, Gordon SC, Patel K, Reau N, Mangia A, Sulkowski M; ASTRAL-2 Investigators; ASTRAL-3 Investigators. Sofosbuvir and Velpatasvir for HCV Genotype 2 and 3 Infection. N Engl J Med. 2015 Dec 31;373(27):2608-17. doi: 10.1056/NEJMoa1512612. Epub 2015 Nov 17. PMID 26575258
- [Background] Younossi ZM, Stepanova M, Sulkowski M, Foster GR, Reau N, Mangia A, Patel K, Brau N, Roberts SK, Afdhal N, Nader F, Henry L, Hunt S. Ribavirin-Free Regimen With Sofosbuvir and Velpatasvir Is Associated With High Efficacy and Improvement of Patient-Reported Outcomes in Patients With Genotypes 2 and 3 Chronic Hepatitis C: Results From Astral-2 and -3 Clinical Trials. Clin Infect Dis. 2016 Oct 15;63(8):1042-1048. doi: 10.1093/cid/ciw496. Epub 2016 Jul 20. PMID 27444413
- [Background] Agarwal K, Castells L, Mullhaupt B, Rosenberg WMC, McNabb B, Arterburn S, Camus G, McNally J, Stamm LM, Brainard DM, Mani Subramanian G, Marino Z, Dufour JF, Forns X. Sofosbuvir/velpatasvir for 12 weeks in genotype 1-4 HCV-infected liver transplant recipients. J Hepatol. 2018 Sep;69(3):603-607. doi: 10.1016/j.jhep.2018.05.039. Epub 2018 Jun 8. PMID 29886154
- [Background] Reau N, Kwo PY, Rhee S, Brown RS Jr, Agarwal K, Angus P, Gane E, Kao JH, Mantry PS, Mutimer D, Reddy KR, Tran TT, Hu YB, Gulati A, Krishnan P, Dumas EO, Porcalla A, Shulman NS, Liu W, Samanta S, Trinh R, Forns X. Glecaprevir/Pibrentasvir Treatment in Liver or Kidney Transplant Patients With Hepatitis C Virus Infection. Hepatology. 2018 Oct;68(4):1298-1307. doi: 10.1002/hep.30046. Epub 2018 Jul 25. PMID 29672891
- [Background] Durand CM, Bowring MG, Brown DM, Chattergoon MA, Massaccesi G, Bair N, Wesson R, Reyad A, Naqvi FF, Ostrander D, Sugarman J, Segev DL, Sulkowski M, Desai NM. Direct-Acting Antiviral Prophylaxis in Kidney Transplantation From Hepatitis C Virus-Infected Donors to Noninfected Recipients: An Open-Label Nonrandomized Trial. Ann Intern Med. 2018 Apr 17;168(8):533-540. doi: 10.7326/M17-2871. Epub 2018 Mar 6. PMID 29507971

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 54 Kidney transplant candidates were enrolled and listed on the Deceased Donor Kidney Wait-list to receive hepatitis C virus (HCV) viremic kidneys
Pre-assignment Details: In total 18 patients were removed from the study: 9 participants received hepatitis C virus nucleic antigen test (HCV NAT) negative kidney transplants, 8 participants were removed from the kidney transplant deceased waiting-list, and 1 participant died prior to receiving kidney transplant
Period: Overall Study
Arm/Group | Intervention Group
Started | 36
Completed | 30
Not Completed | 6
Not completed — Removed from study due to reaching the study target of 30 transplant from hepatitis C viremic donors | 6

BASELINE CHARACTERISTICS:
Arm/Group | Intervention Group
Number analyzed (Participants) | 30
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 59 [51 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 25
  More than one race | 0
  Unknown or Not Reported | 0
Primary cause of end stage kidney diseaes [Count of Participants; unit: Participants]
  Diabetes Mellitus | 11
  Hypertension | 4
  Adult polycystic kidney disease | 7
  Immunoglobin (IgA) nephropathy | 3
  Others | 5
Time on dialysis prior to transplant [Median (Inter-Quartile Range); unit: months] | 12 [8 to 24]
Donor (D) -Recipient (R) Cytomegalovirus (CMV) status [Count of Participants; unit: Participants]
  Cytomegalovirus (CMV) Donor (D)+/ Recipient (R-) | 10
  CMV D+/R+ | 3
  CMV D-/R+ | 10
  CMV D-/R- | 7
Insurance type [Count of Participants; unit: Participants]
  Public, Medicaid | 2
  Public, Medicare | 18
  Private | 10
Pre-Transplant Calculated Panel Reactive Antibody (cPRA) % [Median (Inter-Quartile Range); unit: percent] | 0 [0 to 10]

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Undetectable Hepatitis C Virus (HCV) Polymerase Chain Reaction (PCR) at 12 Weeks After Completion of HCV Treatment
Description: Proportion of patients with undetectable hepatitis C virus (HCV) polymerase chain reaction (PCR) at 12 weeks after completion of HCV treatment was to test the efficacy of the treatment.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group
Number analyzed (Participants) | 30
Participants | 28

2. Primary Outcome: Elevation in Liver Enzyme >5 Times the Upper Limits, Development of Acute Cholestatic Hepatitis , or Intolerance to Direct Acting Antiviral Therapies
Description: Elevation in liver enzyme >5 times the upper limits, development of acute cholestatic hepatitis , or intolerance to Direct acting antiviral therapies was to test the safety of utilizing HepC positive kidneys for transplant.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group
Number analyzed (Participants) | 30
Participants
  Liver enzyme elevation > 5 times upper limit | 2
  Acute cholestatic hepatitis | 0
  Medication intolerance to Direct Acting Antiviral | 0
  No significant adverse effect reported | 28

3. Secondary Outcome: Estimated Glomerular Filtration Rate (eGFR) at 6 and 12 Months Post-transplant
Description: Estimated glomerular filtration rate (eGFR) at 6 and 12 months post-transplant was to test the safety of utilizing of HepC positive kidneys.
Time Frame: 6 and 12 months
Measure: Median (Inter-Quartile Range); unit: ml/min/1.73m^2
Arm/Group | Intervention Group
Number analyzed (Participants) | 30
ml/min/1.73m^2
  eGFR at 6 months | 54 [41 to 68]
  eGFR at 12 months | 46 [40 to 63]

4. Secondary Outcome: Patient's Survival at 6 and 12 Months
Description: Patient's survival at 6 and 12 months measuring safety of utilizing of HepC positive kidneys.
Time Frame: 6 and 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group
Number analyzed (Participants) | 30
Participants
  6 months patient survival | 30
  12 months patient survival | 30

5. Secondary Outcome: Graft Survival at 6 and 12 Months
Description: Graft survival at 6 and 12 months measuring safety of utilizing HepC positive kidneys.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group
Number analyzed (Participants) | 30
Participants
  6 months graft survival | 30
  12 months graft survival | 30

ADVERSE EVENTS:
Time Frame: 25 months
Arm/Group | Intervention Group
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 2/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Group (N=30)
Liver enzyme elevation (Hepatobiliary disorders) | 2 (2) — liver enzyme elevation > 5 upper normal limit occurred in two patients. one patient prior to initiation of direct acting antiviral therapy, one patient during recurrence of HCV viremia in the setting of resistant mutation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-01-14): https://cdn.clinicaltrials.gov/large-docs/07/NCT03801707/Prot_SAP_ICF_001.pdf